CLINICAL TRIAL: NCT00357422
Title: Prospective Randomized Trial of the Effective Therapy for Small, Solitary HCC Comparing Operation and Percutaneous Ethanol Injection Therapy
Brief Title: Comparison Study of Operation and PEIT for Small, Solitary Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-2007-006
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC, operation, percutaneous ethanol injection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Active Comparator)
  Interventions: Procedure: Operation
- local therapy (Active Comparator)
  Interventions: Procedure: Percutaneous ethanol injection therapy

INTERVENTIONS:
Procedure: Operation — No drug needed
  Other Names: surgery
  Arms: surgery
Procedure: Percutaneous ethanol injection therapy — 99% ethanol, 2-4cc per one session, two to three sessions per single procedure for one week
  Other Names: PEIT
  Arms: local therapy

SUMMARY:
The purpose of this study is to choose the preferred treatment modality for solitary, small hepatocellular carcinoma.

DETAILED DESCRIPTION:
To compare the below things between operation group and percutaneous ethanol injection therapy (PEIT) group:

1. Survival

   * 5 year overall survival rate
   * Disease free survival rate
2. Recurrence

   * Cumulative recurrence rate

ELIGIBILITY:
Inclusion Criteria:

* The evidences of hepatitis B virus (HBV)&/or hepatitis C virus (HCV) infection or liver cirrhosis
* Single tumor nodule with Child-Pugh classification A (serum albumin ≥ 3.2 g/dL)
* The maximal, longest diameter of tumor mass measured by CT finding should be less than 2 cm
* Only for the newly detected HCCs which were not treated before
* It should be compatible with the typical finding of hepatocellular carcinomas (HCCs) radiologically (MD CT or dynamic MRI)
* Without portal hypertension

Exclusion Criteria:

* In case of hepatic vein or portal vein invasion radiologically (CT or MRI)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
overall survival rate | 5 year

SECONDARY OUTCOMES:
disease free survival rate and recurrence rate | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: J H Yoon, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul NUH, Seoul, Chongno-gu, South Korea